CLINICAL TRIAL: NCT05383807
Title: Evaluating the Effectiveness of a Social Media-Based Intervention ("Warna-Warni Waktu") to Reduce Body Dissatisfaction Among Young Indonesian Women: Parallel Randomized Controlled Trial
Brief Title: Evaluating a Social Media-Based Intervention to Reduce Body Dissatisfaction Among Young Indonesian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry); University of Hawaii (Other); Indonesia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRR1-10.2196/33596
Record Dates: First submitted 2022-03-29; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-03

CONDITIONS: Body Image
Keywords: body dissatisfaction; body satisfaction; positive body image

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The datasets given to the statistician will be masked to the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warna-Warni Waktu intervention (Experimental): Participants in this condition are asked to view six, approximately five-minute videos (each with a number of associated short, interactive reinforcer activities), at a pace of one video per day, for 6 days.
  Interventions: Behavioral: Warna-Warni Waktu
- Waitlist control condition (No Intervention): These participants are not contacted during the intervention timeframe.

INTERVENTIONS:
Behavioral: Warna-Warni Waktu — Six videos and eighteen reinforcer activities
  Arms: Warna-Warni Waktu intervention

SUMMARY:
The researchers conduct a randomised controlled trial to evaluate a social media-based intervention aimed at reducing body dissatisfaction among young Indonesian women between 15 and 19 years old.The intervention (titled Warna-Warni Waktu) consists of six sequential videos that tell a fictional story of a typical Indonesian young woman. The videos address known risk factors for body dissatisfaction and include evidence-based techniques to mitigate body dissatisfaction. In addition, the intervention encompasses 18 short online activities intended to encourage participants to think critically about the messages learnt in the videos and practice applying the lessons in real life.

The primary aim is to evaluate the short-term (immediate and four-week post) impact of the intervention on young Indonesian women. The primary outcome is trait body dissatisfaction. Secondary outcomes include internalisation of societal appearance ideals, mood, and skin shade satisfaction.

The second aim is to evaluate the effectiveness of the videos individually on eliciting state-based improvements (i.e., improvements in the moment) in body dissatisfaction and mood. This will be a within-group design, whereby only participants in the intervention condition complete single-item measures of body dissatisfaction and mood immediately before and after watching each episode. Further exploratory analyses are also planned.

Approximately 2000 young Indonesian women are recruited for this research project.

The study's hypotheses are as follows:

1. Participants randomised to the intervention condition experience improved body satisfaction, mood, and skin shade satisfaction, and reduced internalisation of appearance ideals at post-intervention (1 day following the intervention), and 1 month follow-up, relative to the waitlist control condition.
2. Each video in the Warna-Warni Waktu series elicits immediate state-based improvements in body satisfaction and mood.
3. Greater engagement and adherence in the Warna-Warni Waktu intervention results in greater body satisfaction, mood, skin shade satisfaction, and reduced internalisation of appearance ideals. This analysis is exploratory in nature, depending on participants' engagement and adherence in the intervention during the trial.

DETAILED DESCRIPTION:
Background

There is a need for culturally-relevant, accessible, and scalable prevention efforts to reduce body dissatisfaction and improve positive body image among Indonesian girls. Currently, no body image interventions for this population exist.

Recruitment

Participants are recruited using a local research agency's database of previous research participants.

Previous participants over the age of 40 are contacted via telephone and screened regarding having a daughter within the eligible age range. If the respondent has more than one daughter in the age range, only one is eligible. If the respondent does not have a daughter between 15 and 19 years of age, the recruiter enquires if the respondent knows another family with a daughter of this age. If so, the recruiter requests the telephone number of that family in order to make contact. Only one phone number is requested per call.

Should an eligible daughter be 15-17 years old, the recruiter reads the parental information sheet to the parent. Parents are then requested to provide verbal consent for the daughter's participation, as well as verification of the parents' identity and daughter's age. Parents then answer questions relating to the family's socio-economic status before the recruiter requests to speak to the daughter. If the daughter is not present, the recruiter requests a call back. The daughter is then screened for eligibility and informed verbal assent obtained. Following a successful call, the parental information sheet is sent to the parent via WhatsApp, and written informed parental consent obtained.

Should an eligible daughter be aged 18 or 19 years old, a similar pattern of communication occurs. Parents verify the age of the parents and the daughter, and respond to questions regarding the family's socio-economic status. Rather than parents providing informed verbal and written consent, this is completed by the daughters, in the same manner with which it is completed by parents of those aged 15-17 years. Verification of identities and ages is achieved through video calls via the presentation of a National ID card and family registration card.

Intervention

The intervention, Warna-Warni Waktu (translation to English: Colourful Time Travel), was developed over a 20-month period, from October 2019 to May 2021. In addition to the close collaboration amongst body image academics, creative agencies, social media specialists, not-for-profit organisations, as well as industry funders, development involved three rounds of feedback from the intervention's target audience.

The narrative story told in the six-video series is based on the concept of time travel so as to convey the additive impact of body image concerns to young people. A combination of both animated characters and real people are used.

Four risk factors for the development of body image concerns are relevant, as identified by the researchers: 1) social media and influencers 2) appearance-based comparisons 3) appearance-based teasing, and 4) body talk. Each of these risk factors are targeted in videos two through five, with videos one and six being the introductory and concluding videos. Each video is four to five minutes in length. A number of change techniques (including those based upon psychoeducation and media literacy) are embedded within the videos.

Each video is accompanied by one to five short interactive activities, designed to elicit cognitive dissonance. Research consistently shows body image interventions that are interactive generate the most positive outcomes.

Procedure

All participants enter the study (i.e., complete the baseline assessment questionnaire) on the same day (Day 1). Participants receive a data package a day prior to this from the research agency to ensure participants have ample mobile phone data to allow participation in the study. A link to the baseline assessment, hosted on Qualtrics (Qualtrics, Provo, UT), is sent to participants via WhatsApp, along with a unique participant identification number (PIN). Participants are requested to enter the PIN on the first page of the baseline survey, in order to match participant responses over time. Participants have 24 hours to complete the baseline assessment; participants that have not completed the baseline assessment within the first 8 hours are sent a reminder message. Following the 24-hour window, participants who have completed the baseline assessment are randomised into one of the two conditions. Participants are alerted on Day 2 to what happens next, depending on which condition each has been randomised. Participants randomised to the intervention condition are informed to expect a series of links to be sent over the following six days. Participants in the control condition are informed that contact will be made again in one weeks' time to complete a second assessment.

On the third day (Day 3), participants in the intervention condition are sent the unique PIN and a link to the first video in the intervention. Again, participants are requested to enter the unique PIN on the first page of the link. Before watching video one in the Warna-Warni Waktu series, participants complete state measures of body satisfaction and affect. State measures of body satisfaction and affect are asked again, immediately after the video. Next, participants are presented with the reinforcer activities for video one to complete. This process is repeated on Days 4-8, for videos two-six.

On Day 9 of the study, participants in both conditions are sent a link to complete the second assessment. As with the baseline assessment, participants are given 24 hours to complete this assessment, with reminder messages sent to non-completers after the first eight hours. The same process is executed for the third and final assessment, one month later on Day 37.

Following the third assessment, all participants are debriefed on the study aims and provided with additional sources of mental health support, as well as a certificate of participation. Those in the waitlist control condition are provided with a link to the Warna-Warni Waktu video series to watch, if desired.

ELIGIBILITY:
Inclusion Criteria:

* identifying as a girl
* aged between 15 and 19 years old
* own their own mobile phone
* access Facebook or Instagram daily.

Exclusion Criteria:

* follow the Girl Effect brand ('Springster') on any social media site
* have ever accessed the Springster website
* if under 18 years of age, do not have the written consent from a parent or guardian.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Eligibility is determined based on an individual identifying as female.
Enrollment: 2000 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Change in body esteem | baseline; post-intervention (1 day after the intervention is complete); follow-up (4 weeks later)
  Body esteem (body satisfaction) is assessed using the Body Esteem Scale for Adolescents & Adults (Mendelson, Mendelson & White, 2001), newly validated among Indonesian adolescents prior to the trial. Once the appropriate items are reverse coded, scores on all items are averaged; with higher scores indicating higher body esteem.

SECONDARY OUTCOMES:
Change in internalisation of societal appearance ideals | baseline; post-intervention (1 day after the intervention is complete); follow-up (4 weeks later)
  Internalisation of societal appearance ideals is assessed using The Sociocultural Attitudes Towards Appearance Questionnaire-3 (SATAQ-3): General Subscale (Thompson, van de Berg, Roehrig, Guarda, & Heinberg, 2004), newly validated among Indonesian adolescents prior to the trial. Scores are averaged, with higher scores indicating higher internalisation.
Change in mood | baseline; post-intervention (1 day after the intervention is complete); follow-up (4 weeks later)
  Positive and negative mood is measured using the Positive and Negative Affect Schedule for Children (Laurent, Catanzaro, Joiner, Rudolph, Potter, Lambert, Osborne, & Gathright, 1999), newly validated among Indonesian adolescents prior to the trial. Scores on each subscale are averaged; with higher scores indicating greater negative affect and positive affect respectively.
Change in skin shade satisfaction | baseline; post-intervention (1 day after the intervention is complete); follow-up (4 weeks later)
  Single-item, purpose built measure to assess satisfaction with skin shade.
Change in state body satisfaction | Immediately before and after watching each of the six intervention videos.
  State body satisfaction is measured using a 101-point visual analogue scale (Heinberg & Thompson, 1995)
Change in state mood | Immediately before and after watching each of the six intervention videos.
  State mood is measured using a 101-point visual analogue scale (Heinberg & Thompson, 1995)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Garbett, MSc, Principal Investigator — University of the West of England
Locations (1):
- University of the West of England, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garbett KM, Haywood S, Craddock N, Gentili C, Nasution K, Saraswati LA, Medise BE, White P, Diedrichs PC, Williamson H. Evaluating the Efficacy of a Social Media-Based Intervention (Warna-Warni Waktu) to Improve Body Image Among Young Indonesian Women: Parallel Randomized Controlled Trial. J Med Internet Res. 2023 Apr 3;25:e42499. doi: 10.2196/42499. PMID 37010911